CLINICAL TRIAL: NCT01890772
Title: A Pilot Trial of the Safety and Efficacy of Telaprevir +Peginterferon +Ribavirin +Vitamin D3 Among Treatment-naive Veterans Infected With Genotype 1 Hepatitis C Virus
Brief Title: Vitamin D + Telaprevir + Peginterferon + Ribavirin for of Hepatitis C Genotype 1
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Timothy Morgan, MD (Other)
Collaborators: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor-Investigator, Timothy Morgan, MD, Chief, Hepatology, Southern California Institute for Research and Education
Organization: Southern California Institute for Research and Education (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1217
Record Dates: First submitted 2013-05-31; First posted 2013-07-02 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2014-05

CONDITIONS: Hepatitis C
Keywords: Hepatitis C Genotype 1; Vitamin D; treatment-naive
MeSH Terms: conditions — Hepatitis C | interventions — telaprevir; peginterferon alfa-2a; Ribavirin; Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- VitD+telaprevir+peginterferon+ribavirin (Active Comparator): Participants randomized to the treatment group will receive 5,000IU/day of vitamin D3 during the lead-in phase. When the serum 25(OH)D level is ≥35ng/ml the participant will begin telaprevir + vitamin D3 (15,000IU/week) + peginterferon alfa-2a (180ug/week) + weight based ribavirin treatment.
  Interventions: Drug: Telaprevir; Drug: Peginterferon alfa-2a; Drug: Ribavirin; Dietary Supplement: Vitamin D
- Telaprevir + Peginterferon + Ribavirin (Active Comparator): Participants randomized to the control group immediately begin treatment with telaprevir + 180ug of peginterferon alfa-2a (Pegasys) per week and either weight based ribavirin.
  Interventions: Drug: Telaprevir; Drug: Peginterferon alfa-2a; Drug: Ribavirin

INTERVENTIONS:
Drug: Telaprevir
  Other Names: Incivek
Drug: Peginterferon alfa-2a
  Other Names: Pegasys
Drug: Ribavirin
Dietary Supplement: Vitamin D
  Arms: VitD+telaprevir+peginterferon+ribavirin

SUMMARY:
This study is for people who have been diagnosed with chronic hepatitis C, specifically those who have a certain type of the virus, genotype 1, and who have not yet received treatment for hepatitis C. This pilot study is designed to test whether the addition of vitamin D, to the three drugs (Incivek (telaprevir), Pegasys (peginterferon alfa-2a), and ribavirin) that are approved by the Food and Drug Administration (FDA) for the treatment of hepatitis C, can help eliminate the HCV from the body. Currently, doctors are unsure if the addition of vitamin D to prescribed hepatitis C therapy will have any effects on how the body clears the virus.

Once enrolled, participants will be randomly assigned (like flipping a coin) to receive telaprevir + peginterferon alfa-2a + ribavirin + vitamin D3 (treatment group) or telaprevir + peginterferon alfa-2a + ribavirin (control group). A total of 80 participants, of all races/ethnicities, will be included in this study, at 5 to 10 VA hospital study sites (10 - 20 participants/site).

Participants assigned to the treatment group will begin a lead-in phase where they will receive 5,000 IU of vitamin D3 per day. Every two weeks during the lead-in phase, participants will be tested to determine the Vitamin D level in their blood, as well as other tests, including HCV RNA (to determine the amount of virus present) and calcium levels. Once an adequate level of Vitamin D is detected in participants' blood, participants will begin treatment with telaprevir + peginterferon alfa-2a + ribavirin + vitamin D3 (15,000 IU/week) for 12 weeks.

Participants randomized to the control group will immediately begin treatment with telaprevir + peginterferon alfa-2a + ribavirin for 12 weeks. At the end of Week 12 the participants' involvement in the study will be complete.

Adverse events and effects of vitamin D3 will be obtained by assessing participants' medical history, physical examination, and blood tests at clinic visits. HCV RNA will be assessed at Screening, Day 1, Week 2, 4, 8 and 12.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Hepatitis C genotype 1 infection
* Treatment naïve
* Age >18 years
* Agree to genetic testing

Exclusion Criteria:

* Liver disease other than from hepatitis C
* HCV infection with mixed genotypes
* Decompensated liver disease
* AFP>100ng/ml.
* Known HIV infection
* Serum 25(OH)D less than 12ng/ml or greater than 30ng/ml
* Regular vitamin D supplement use
* Regular calcium supplement use
* Refusal to abstain from vitamin D supplementation
* Current or past history of kidney stones
* Current use of any of the prohibited medications listed in section 5.5 and the INCIVEK® package insert.
* Need for therapeutic vitamin D or calcium (e.g. treatment for osteoporosis, osteomalacia, hyperparathyroidism etc.), in the opinion of the investigator
* Significant substance abuse within the past 6 months,
* Suicidal attempt in the past 10 years or suicidal ideation in past 3 months, or any other psychiatric condition that the investigator deems would make a subject unsuited for treatment with peginterferon or ribavirin.
* Confirmed or suspected malignancy, or history of malignancy within the past 3 years (except treated basal cell carcinoma of the skin or in situ carcinoma of the uterine cervix)
* Any autoimmune disease not easily controlled (in the opinion of the investigator)
* Any condition resulting in malabsorption (
* Poorly controlled thyroid disorder, or diabetes mellitus (HbA1c > 9)
* Glomerular diseases (e.g., glomerulosclerosis or glomerulonephritis) associated with a serum creatinine >1.5 times the upper limit of normal
* Current or history of any clinically significant cardiac abnormalities/dysfunction (eg, angina, congestive heart failure, myocardial infarction, pulmonary hypertension, complex congenital heart disease, cardiomyopathy, significant arrhythmia) including current uncontrolled hypertension or history of use of antianginal agents for cardiac conditions (Inclusion will be considered if clearance by a cardiologist is obtained.)
* Receipt of an investigational drug within the past 30 days
* Females who have a positive pregnancy test at the time of screening, are breastfeeding or who anticipate pregnancy within the next 18 months, or men with pregnant partners
* Lack of agreement from subject to use two forms of acceptable contraception
* History or other evidence of any significant illness which, in the opinion of the investigator, would make the patient, unsuitable for the study
* Laboratory Exclusions

Hemoglobin: <12gm/dl male or female

Neutrophil: <1,200/mm3

Platelets: <90,000/mm3

INR: >1.5

Albumin: <3.2gm/dl

Total Bilirubin: >2.0mg/dl

HbA1c: >9.5%

Serum Creatinine: >1.5 times the upper limit of normal

Serum Calcium Within local laboratory normal range

Parathyroid hormone (PTH) <10 or >55 pg/mL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-08; Primary Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
HCV RNA | 4 weeks
  Hepatitis C virus Ribonucleic Acid identifies the presence of Hepatitis C in the blood

SECONDARY OUTCOMES:
adverse event profile | 12 weeks
  Cumulative record of unanticipated or unintended medical occurrences, not necessarily related to the study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy R Morgan, MD, Principal Investigator — Veterans Affairs Long Beach Healthcare
Locations (4):
- United States (4):
  - VA Long Beach Healthcare System, Long Beach, California
  - Minneapolis VAHCS, Minneapolis, Minnesota
  - Kansas City VA Medical Center, Kansas City, Missouri
  - Philadelphia VA Medical Center, Philadelphia, Pennsylvania